CLINICAL TRIAL: NCT05767255
Title: Risk of Hypoglycemia in the Transition From Inpatient to Outpatient Setting. Comparative Study of Basal-bolus Insulin Versus Basal Insulin Plus GLP-1 Analogue
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/145
Record Dates: First submitted 2023-02-16; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2 Treated With Insulin
Keywords: IDegLira; Type 2 diabetes mellitus; Glycemic; Diabetes medications.
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized 1:1 to continue the basal bolus ( insulin glargine and aspart ) or IDegLira ( insulin glargine and aspart ) or IDegLira ) on an outpatient basis by means of a system of random number generation through a mobile application ( Random Number Generator ) that will be centralized ( by a member of the independent group ) and to which the rest of the investigators will not have access.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- basal group bolus (Active Comparator): * Insulin Glargine required on an in-hospital basis
  * Insulin Aspart required on an in-hospital basis
  Interventions: Drug: Insulin Glargine - Insulin Aspart
- insulin degludec + liraglutide ( ideglira) (Experimental): 16 Units once a day
  Interventions: Drug: insulin degludec + liraglutide

INTERVENTIONS:
Drug: insulin degludec + liraglutide — The association of insulin degludec with liraglutide in the same device (IDegLira) is a potent and safe drug that reduces the risk of hypoglycemia.
  Other Names: ideglira
  Arms: insulin degludec + liraglutide ( ideglira)
Drug: Insulin Glargine - Insulin Aspart — The insulin dose of the basal group will be adjusted according to the blood glucose reports presented by the patients.
  Arms: basal group bolus

SUMMARY:
The association of insulin degludec with liraglutide in the same device (IDegLira) is a potent but at the same time safe drug that reduces the risk of hypoglycemia when compared to a basal or basal-bolus insulin schedule.

The DUAL (Dual Action of Liraglutide and Insulin Degludec) studies are the pivotal studies of this combination. Specifically, the DUAL VII study has demonstrated that ideglira is a non-inferior drug in terms of glycemic control versus a basal-bolus schedule in patients in the outpatient setting who have failed basal insulin.

Although the basal-bolus insulin plus correction schedule is frequently used in hospitalized patients with hyperglycemia, outpatient management with a complex insulin schedule creates challenges that are difficult to mitigate due to limited time for patient education during an acute illness and limited access to the physician responsible for post-discharge diabetes management.

The use of IDegLira has not been evaluated in clinical studies in the hospital discharge setting where the authors believe it has great potential because it offers similar potency to the basal-bolus scheme but with greater safety with respect to hypoglycemia and less complexity for the patient because it is associated with fewer applications and less need for capillary self-monitoring.

For this reason, in the hospital-home transition scenario, ideglira therapy in patients with poor metabolic control and requiring intensification therapy is proposed as an alternative to the basal-bolus scheme.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (DM 2) is a chronic non-communicable metabolic disease characterized by progressive deterioration of beta cell functionality, which associated with the presence of insulin resistance results in persistent elevations of plasma glucose or hyperglycemia. The objectives of its treatment are to prevent or delay complications and optimize quality of life.

The American Diabetes Association (ADA) consensus report "Standards of Medical Care in Diabetes-2021" recommends a patient-centered approach to choosing appropriate pharmacologic treatment of glycemia. This includes consideration of key patient factors: 1) important comorbidities, such as atherosclerotic cardiovascular disease, high-risk indicators of cardiovascular, chronic kidney disease, and heart failure, 2) risk of hypoglycemia, 3) effects on body weight, 4) side effects, 5) cost, and 6) patient preferences.

With these considerations in mind, drug therapy should be initiated in conjunction with a lifestyle modification consultation focused on diet and physical activity. Considering the progressive nature of the disease, monotherapy only achieves glycemic control for a few years and treatment intensification is required as the disease progresses, however, therapeutic inertia leads to delayed intensification in diabetic patients who are not at glycemic control goals, mainly when it comes to the use of injectable therapies such as insulins.

In recent years, two combinations of basal insulin with GLP-1 analog received regulatory approval from the European Medicines Agency and the U.S. Food and Drug Administration Agency. These therapeutic strategies are fixed ratio combinations of insulin degludec U100 and liraglutide (IDegLira); and insulin glargine U100 and lixisenatide (IGlarLixi). Both options demonstrated non-inferiority or superiority in reducing (Hb1Ac) levels in terms of glycemic control compared to their individual components in monotherapy, in the DUAL I study for IDegLira and in the LixiLan-O study for IGlarLixi .

Clinical trials supporting the efficacy and safety of IDegLira in the outpatient setting include DUAL (Dual Action of Liraglutide and Insulin Degludec in Type 2 Diabetes. On the other hand, there are authors who propose considering the use of IDegLira as the first injectable therapy in type 2 diabetic patients and as a therapeutic alternative in those who do not reach glycemic control goals with pharmacological treatment including monotherapy with GLP1 analogues, basal insulin or therapy with multiple doses of insulin in patients with recurrent hypoglycemia.

Considering the above, injectable therapy combined with IDegLira is proposed as an alternative for therapeutic intensification in patients with uncontrolled DM 2, since it has demonstrated efficacy and safety in the management of this pathology, achieving adequate glycemic control while leading to weight loss, lower rates of hypoglycemia and savings in insulin doses, in addition to providing a simple application scheme compared to the basal-bolus scheme.

In patients with DM 2, hospitalization represents an important change in medication: most consensus and guidelines propose the use of insulin therapy for glycemic control during hospital stay.

However, therapy at the time of hospital discharge should be adjusted and reconciled with the use of other non-insulin diabetes medications.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with a diagnosis of type 2 diabetes mellitus who have received basal-bolus insulin during hospitalization and who, at the time of hospital discharge, are considered necessary to continue this scheme (basal-bolus).

Exclusion Criteria:

* Patient with diagnosis or suspicion of DM1.
* Inability of the patient or family member to continue injectable therapy at home.
* CKD with GFR < 15 ml/minute by CKD EPI.
* History of chronic or acute pancreatitis in the last 3 months.
* History of personal or family history of medullary thyroid cancer.
* History of hypersensitivity to any of the components of the IdegLira combination.
* Women in pregnancy, breastfeeding or absence of hormonal contraception.
* Management for obesity with GLP1 receptor agonist.
* Previous management with basal bolus scheme with total daily dose of insulin (DDT) greater than 70 U/day.
* Patients with hyperglycemia associated with steroids.
* Patients who are insulin users prior to current hospitalization and have an in-hospital HbA1c greater than 11%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
To compare the percentage of hypoglycemia | 4 weeks
  To compare the percentage of patients presenting at least one episode of hypoglycemia (defined as one or more episodes of hypoglycemia below 54 mg/ dL for more than 20 minutes by continuous flash glucose monitoring), between the basal bolus group and the degludec/liraglutide (ideglira) group in the first four weeks after hospital discharge.

SECONDARY OUTCOMES:
Compare episodes of severe hypoglycemia | 4 weeks
  To compare episodes of severe hypoglycemia between the two groups; defined as episodes with altered state of consciousness or requiring assistance from another person to make corrective decisions.
Compare the metrics of glycemic control | 4 weeks
  To compare the metrics of glycemic control (time in range 70-180 mg/dL, time above range 180 mg/dL, time above 250 mg/dL , GMI, coefficient of variation ) of the two groups.
Compare the incidence density of hypoglycemia | 4 weeks
  To compare the incidence density of hypoglycemia defined as the number of hypoglycemia events (readings below 54 mg/ dL for more than 20 minutes by continuous flash glucose monitoring) in each intervention group.
compare the percentage of patients without episodes of hypoglycemia | 4 weeks
  To compare the percentage of patients achieving a time in range greater than 70% without episodes of hypoglycemia in each intervention group.
HbA1c change | 4 weeks
  To evaluate the efficacy of the schemes according to Hbac1 metrics before randomization.
To assess whether there is a difference in body weight | 4 weeks
  To assess whether there is a difference in body weight change according to treatment allocation arm.
Evaluate associated adverse effects | 4 weeks
  Evaluate and compare associated adverse effects such as: nausea, emesis, abdominal distension, diarrhea, constipation, epigastric pain, early satiety, postprandial fullness, weight gain, acute pancreatitis, symptomatic cholelithiasis, diabetic ketoacidosis, hyperosmolar state (see attached operational definitions).They will be evaluated by means of the CTCAE manual version 5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Gomez-Medina AM, Henao-Carillo DC, Villamil-Castaneda LP, Gomez-Quesada Y, Munoz-Velandia OM, Yepes CA, Chaim SN, Pertuz-Noriega CE, Aschner P. Insulin DEgludec/LIraglutide versus multiple daily insulin injections in the transition from hospital to outpatient management assessed by continuous glucose monitoring: the DELI transition trial. Diabetologia. 2025 Sep;68(9):1899-1907. doi: 10.1007/s00125-025-06446-y. Epub 2025 Aug 4. PMID 40760249